CLINICAL TRIAL: NCT00344370
Title: Double-Blind, Follow-On Study of Pitavastatin (4 mg) Versus Atorvastatin (20 mg and 40 mg), With a Single-Blind Extension of Treatment, in Patients With Type II Diabetes Mellitus and Combined Dyslipidemia
Brief Title: Follow-On Study of Pitavastatin Versus Atorvastatin in Patients With Type II Diabetes Mellitus and Combined Dyslipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kowa Research Europe (Industry)
Responsible Party: Dragos Budinski, MD, Kowa Research Europe
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NK-104-310
Record Dates: First submitted 2006-06-23; First posted 2006-06-26 (Estimated); Results first posted 2010-01-18 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-01

CONDITIONS: Type II Diabetes Mellitus; Dyslipidemia
Keywords: Pitavastatin; Type II Diabetes Mellitus; Combined Dyslipidemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Dyslipidemias | interventions — pitavastatin; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pitavastatin (Experimental): Pitavastatin 4 mg QD
  Interventions: Drug: Pitavastatin
- Atorvastatin (Active Comparator): Atorvastatin 40 mg
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Pitavastatin — Pitavastatin 4 mg QD
  Other Names: Livalo
  Arms: Pitavastatin
Drug: Atorvastatin — Atorvastatin 40 mg
  Other Names: Lipitor
  Arms: Atorvastatin

SUMMARY:
This is a sixteen-week double-blind active-controlled follow-on and 28-week single-blind extension study for patients who participated in study NK-104-305.

ELIGIBILITY:
Inclusion Criteria:

* Type II diabetes mellitus
* Combined dyslipidemia
* Completed NK-104-305 (NCT00309751)

Exclusion Criteria:

* Withdrawal from NK-104-305 (NCT00309751)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2006-08; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dragos Budinski, MD, Study Director — Kowa Research Europe (KRE)
Locations (35):
- Denmark (3):
  - CCBR Aalborg, Aalborg
  - CCBR A/S, Vejle
  - CCBR Vejle, Vejle
- Germany (5):
  - Gemeinschaftspraxis am Bahnhof, Berlin-Spandau
  - Pharmakologisches Studienzentum Chemnitz, Chemnitz
  - Internistische Diabetische Schwerpunktpraxis Dr., Frankfurt am Main
  - Internistische Gemeinschaftspraxis, Mainz
  - Gemeinschaftspraxis Dr. Senftleber, Dr. Kohler, Messkirch
- India (5):
  - Bhagwan Mahaveer Jain Heart Centre, Bangalore
  - Sri Ramachandra Medical College Hospital, Chennai
  - Apollo Hospitals, Hyderabaad
  - CARE Group of Hospitals, Hyderabaad
  - PD Hinduja Hospital, Mumbai
- Netherlands (8):
  - Andromed Breda, Breda
  - Andromed Eindhoven, Eindhoven
  - Andromed Noord, Groningen
  - Andromed Leiden, Leiden
  - Andromed Nijmegen, Nijmegen
  - Andromed Rotterdam, Rotterdam
  - Andromed Oost, Velp
  - Andromed Zoetermeer, Zoetermeer
- Poland (10):
  - Podlaski Osrodek Kardiologii, Bialystok
  - NZOZ GCP Dobra Praktyka Lekaska, Gruziadz
  - NZOZ Terapia Optima, Katowice
  - NZOZ Centrum, Poradnia Kardiologiczna, Siedlce
  - Spec. Gab. Lek. Internistyczno-Kardiologicznly, Tarnów
  - Woj.Szp.Spec.Nr 1 im. Prof. J. Gasinskiego, Tychy
  - Instytut Zywnosci i Zywienia, Warsaw
  - Lecznica PROSEN SMO, Warsaw
  - Szpital Wolski,im. Dr A. Gostynskiej, Warsaw
  - NZOZ Esculap, Przychodnia Lekary Rodzinnych, Łosice
- United Kingdom (4):
  - Synexus Reading Clinical Research Centre, Berkshire
  - Synexus Lancashire Clinical Research Centre, Lancashire
  - Synexus Merseyside Clinical Research Centre, Liverpool
  - Synexus Manchester Clinical Research Centre, Manchester

RESULTS

PARTICIPANT FLOW:
Groups:
- Pitavastatin 4 mg: Pitavastatin 4 mg once daily
- Atorvastatin 40 mg: Atorvastatin 40 mg once daily
Period: Overall Study
Arm/Group | Pitavastatin 4 mg | Atorvastatin 40 mg
Started | 143 | 71
Completed | 128 | 68
Not Completed | 15 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pitavastatin 4 mg | Atorvastatin 40 mg | Total
Number analyzed (Participants) | 143 | 71 | 214
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 95 | 46 | 141
  >=65 years | 48 | 25 | 73
Age Continuous [Mean (Standard Deviation); unit: years] | 59.3 (9.83) | 60.0 (9.21) | 59.5 (9.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 30 | 98
  Male | 75 | 41 | 116

OUTCOME MEASURES:

1. Primary Outcome: NCEP LDL-C Target Attainment
Description: Number of patients attaining National Cholesterol Education Program (NCEP) LDL-C target at 44 weeks. According to NCEP criteria the target LDL-C is 100 mg/dL for all patients in this study.
Time Frame: 44 weeks
Population: The efficacy population is defined as all patients who received at least one dose of study drug and who had at least one on-treatment lipid assessment
Measure: Number; unit: Participants
Arm/Group | Pitavastatin 4 mg | Atorvastatin 40 mg
Number analyzed (Participants) | 141 | 71
Participants | 110 | 55

2. Secondary Outcome: Percent Change From Baseline in LDL-C
Description: Percent change from baseline in LDL-C at 44 weeks
Time Frame: Basseline to 44 weeks
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Pitavastatin 4 mg | Atorvastatin 40 mg
Number analyzed (Participants) | 141 | 71
percent change | -40.98 (19.053) | -41.43 (21.159)

ADVERSE EVENTS:
Arm/Group | Pitavastatin 4 mg | Atorvastatin 40 mg
Serious Adverse Events (participants affected / at risk) | 8/143 | 5/71
Other Adverse Events (participants affected / at risk) | 22/143 | 15/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pitavastatin 4 mg (N=143) | Atorvastatin 40 mg (N=71)
Acute coronary syndrome (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 | 0
Abdominal wall abscess (Infections and infestations) | 1 | 0
Bacterial pyelonephritis (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pitavastatin 4 mg (N=143) | Atorvastatin 40 mg (N=71)
Myalgia/myalgia intercostal (Musculoskeletal and connective tissue disorders) | 6 | 5
Naspopharyngitis (Musculoskeletal and connective tissue disorders) | 10 | 2
Arteriosclerosis (Vascular disorders) | 4 | 4
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days